CLINICAL TRIAL: NCT01544504
Title: Exploratory Study of Topical Norepinephrine in Post-Surgical Breast Cancer Patients Receiving Radiotherapy
Brief Title: Exploratory Study of Topical Norepinephrine in Breast Cancer Patients Receiving Radiotherapy
Status: Withdrawn | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: The principal investigator withdrew from the study. The study was withdrawn because a qualified replacement was not available.
Sponsor: ProCertus BioPharm, Inc (Industry)
Collaborators: H. Lee Moffitt Cancer Center and Research Institute (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: PC-6
Record Dates: First submitted 2012-02-15; First posted 2012-03-06 (Estimated); Last update posted 2012-05-28 (Estimated); Status verified 2012-05

CONDITIONS: Radiodermatitis
Keywords: Radiodermatitis; Prevention; Radiotherapy; Breast; Radiation Dermatitis
MeSH Terms: conditions — Radiodermatitis | interventions — Norepinephrine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Norepinephrine (Experimental): Topical norepinephrine
  Interventions: Drug: Norepinephrine

INTERVENTIONS:
Drug: Norepinephrine — Approximately 4.65 mL of a norepinephrine solution (400 mM, 82.3 mg/mL) will be applied topically to the study drug application site prior to each radiotherapy treatment (approximately 25-28 treatments).
  Other Names: Noradrenaline

SUMMARY:
This study, a nonrandomized open-label safety and exploratory study, will evaluate the safety of topical norepinephrine in post-surgical breast cancer patients who are undergoing radiation therapy.

The study will also provide information about whether topical norepinephrine can prevent or decrease the severity of the radiation dermatitis experienced by these patients.

ELIGIBILITY:
Inclusion Criteria:

Subjects must:

1. be ≥ age 18 years of age with a documented pathological diagnosis of Stage Ia (T1, N0, M0), Stage Ib (T0 or 1, N1mic, M0), Stage IIA (T0-T1N1M0, T2N0M0) or Stage IIB (T2N1M0, T3N0M0) infiltrating ductal or lobular carcinoma of the breast or ductal carcinoma in situ (DCIS).
2. be post-surgical patients scheduled to be treated with at least 50 Gy to the whole breast and axilla using standard radiation techniques (an additional 10-16 Gy boost to the lumpectomy region may also be delivered). All radiation treatment is to be delivered based on standard CT planning.
3. be at higher than average risk for radiodermatitis, as evidenced by a separation at the posterior tangent field border of ≥ 24 cm or a bra cup size of C or greater [breast size criterion].
4. have the ability to understand the informed consent document.
5. be able to comply with protocol schedule.
6. have a negative serum pregnancy test (within 7 days prior to starting radiation therapy), if a female of child bearing potential.
7. consent to utilize medically acceptable methods of contraception throughout the study period if of child-bearing potential.

Exclusion Criteria:

Subjects:

1. with unhealed surgical wounds or scars in the study treatment area.
2. with underlying active untreated cardiac disease (e.g. arrhythmia).
3. with generalized skin disorders that have required treatment within the past 6 months.
4. with connective tissue disorders.
5. with rashes, ulcerations, or poorly healed scars in the study drug application area.
6. with a known allergy to norepinephrine.
7. with a known clinically significant abnormal ECG within the past 6 months. If the Principal Investigator feels that the ECG findings are of clinical significance, the patient will excluded or sent for a cardiac consult (insignificant abnormalities such as sinus tachycardia and sinus bradycardia may be allowed at the discretion of the Principal Investigator).
8. receiving MAO inhibitors or antidepressants (triptyline or imipramine types).
9. who are pregnant or breastfeeding.
10. with lymphovascular space invasion on pathology.
11. with dermal lymphatic invasion on pathology.
12. with close proximity of the tumor to the overlying skin within the SDAS (as evidenced by a depth of less than 5 mm on ultrasound or MRI [if performed] and a linear distance of less than 2 cm from the SDAS), or a diagnosis of inflammatory breast cancer.
13. receiving concurrent neoadjuvant or adjuvant chemotherapy for their breast cancer.
14. with previous radiation to the breast to be treated.
15. taking β-blockers.
16. with NCI CTC Version 4.0 grade 2 or higher hypertension at the time of study entry.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2012-03; Primary Completion 2012-05 (Actual); Study Completion 2012-05 (Actual)

PRIMARY OUTCOMES:
Safety of daily topical application of norepinephrine to the radiation field | Safety will be assessed for up to 11 weeks following the start of treatment.
  The primary safety hypothesis is that there will be little or no skin irritation associated with the application of the topical norepinephrine and no systemic effects secondary to transdermal absorption.

SECONDARY OUTCOMES:
Efficacy of daily topical application of norepinephrine to the radiation field | Efficacy will be assessed for up to 11 weeks following the start of treatment..
  The primary efficacy hypothesis is that the portion of the radiation site that is treated with topical norepinephrine immediately prior to daily radiotherapy will have less severe radiation dermatitis than the adjacent untreated portion of the radiation site.

CONTACTS AND LOCATIONS:
Overall Officials: Eleanor Harris, MD, Principal Investigator — H. Lee Moffitt Cancer Center and Research Institute
Locations (1):
- H Lee Moffitt Cancer Center and Research Institute, Tampa, Florida, United States